CLINICAL TRIAL: NCT07100808
Title: Evaluation of Clinical Efficacy of Subepithelial Connective Tissue Graft and Free Gingival Graft De-Epithelialized With Two Different Methods in the Treatment of Gingival Recessions
Brief Title: Evaluation of the Clinical Efficacy of De-Epithelialized Free Gingival Graft in the Treatment of Gingival Recessions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Nazli Zeynep Alpaslan, Associate Professor, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 17.06.2020/14
Record Dates: First submitted 2025-07-03; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Gingival Recessions
Keywords: Laser Therapy; Gingival Recession; autografts
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Subepithelial Connective Tissue Grafts Group (Active Comparator): The single incision technique was used as a guide for harvesting the SCTG from the palatal region. After achieving hemostasis in the palatal area, the incision site was primarily closed using 4-0 silk sutures with a cross-suture technique. The graft, held with guide sutures, was slid beneath the interdental papillae and placed into the tunnel bed. The elevated papillary complex was sutured together with the graft using 5-0 monofilament sutures (Neoplene, polypropylene, Turkey) and secured coronally and over the root surface, covering the graft, using vertical double-cross sutures. The surgical procedure, suturing technique, and sutures used on the recipient site were standardized across all groups.
  Interventions: Procedure: Using the tunnel technique in the treatment of gingival recession
- •Scalpel-based De-epFGG Group (Active Comparator): In this group, the De-epFGG technique recommended by Zucchelli et al. was applied. The epithelial layer on the outer surface of the harvested graft was removed by holding a 15C scalpel (Swann-Morton LTD, Sheffield, England) parallel to the surface. The prepared CTG was then placed in the tunnel bed at the desired position using guide sutures.
  Interventions: Procedure: Using the tunnel technique in the treatment of gingival recession
- Er,Cr:YSGG Laser-based De-epFGG Group (Active Comparator): Before the laser application, patients were asked to wear the necessary protective eyewear. The graft dimensions required for the recipient site were marked on the palatal donor area using a 15C scalpel.
  The donor site was irradiated with a 2780 nm Er,Cr:YSGG laser (WaterLase iPlus; USA Biolase Technology Inc., Irvine, CA), and the de-epithelialization procedure was completed intraorally. The surface layer formed as a result of the laser application was removed using a moist sponge.
  Interventions: Procedure: Using the tunnel technique in the treatment of gingival recession

INTERVENTIONS:
Procedure: Using the tunnel technique in the treatment of gingival recession — Microsurgical periodontal instruments were used during surgical procedures. In this study, specially developed tunnel instruments (Helmunt Zepf, Seitingen-Oberflacht, Germany) were used to mobilize the gingivo-papillary unit and prepare the supraperiosteal tunnel bed. After passing the coronal edge of the alveolar bone with the tunnel instrument placed in the soft tissue, it was advanced towards the apical mucogingival junction with small, circular movements. This procedure was repeated by entering from the sulcus of each tooth. Care was taken to ensure that the prepared flaps were in the same layer and opened towards each other. In the interdental areas, the papillary complex was carefully separated from the periosteum and mobilized in the buccal direction. Thus, mobilization of the entire buccal soft tissue complex was achieved in the coronal direction. After these procedures, it was checked whether the flap covered the recession areas without tension.
  Other Names: Mucogingival surgery

SUMMARY:
The aim of this study is to evaluate the clinical effectiveness of three techniques used in combination with the tunnel method for the treatment of multiple gingival recessions: subepithelial connective tissue graft (SCTG Group), scalpel-de-epithelialized free gingival graft (Scalpel Group), and Erbium, Chromium: Yttrium-Scandium-Gallium-Garnet (Er,Cr:YSGG) laser-de-epithelialized free gingival graft (Laser Group).

DETAILED DESCRIPTION:
Gingival recession is not only one of the most common aesthetic and functional problems of the periodontium, but also one of the most complex conditions in terms of etiology and treatment modalities. Subepithelial connective tissue grafts (SCTG), applied in combination with various techniques, are considered the gold standard in the treatment of gingival recession. In cases where a surgical approach is indicated, coronally advanced flap (CAF) or graft-based subepithelial connective tissue procedures in combination with the tunnel technique (TT) have been reported to be successfully utilized.

The use of de-epithelialized free gingival graft (De-epFGG) as a connective tissue graft (CTG) represents another treatment option for managing gingival recession.

With advancements in laser technology, lasers with various wavelengths are increasingly being used as alternatives to scalpels in numerous intraoral surgical procedures. Considering the advantageous properties of erbium lasers, which are among the most prominent dental lasers, their use has also been demonstrated for preparing recipient sites for free gingival grafts (FGG). There are only a limited number of studies in the literature investigating the combination of De-epithelialized Free Gingival Graft (De-epFGG) with the Tunnel Technique (TT). The aim of this study is to evaluate the clinical effectiveness of SCTG, scalpel-based De-epFGG, and Er,Cr:YSGG laser-based De-epFGG techniques, all applied in combination with the tunnel technique, in the treatment of Miller Class I and II multiple gingival recessions.

The study hypothesis is that the percentage of root coverage achieved using De-epFGG (scalpel and laser methods) would be comparable and that these methods could serve as strong alternatives to SCTG.

ELIGIBILITY:
Inclusion Criteria:

Presence of Miller Class I or II recession defects in at least two adjacent teeth in the maxillary or mandibular arch

* Recession depth ≥ 2 mm
* Recession areas present on intact, caries-free teeth with no restorations

Exclusion Criteria:

* ▪ History of periodontal surgery in the target area within the past 6 months

  * Use of antibiotics within the past 6 months
  * Pregnancy or lactation
  * Presence of Miller Class III or IV gingival recession
  * Recession defects on molar teeth
  * Undergoing orthodontic treatment,
  * Presence of parafunctional habits
  * Individuals with contraindications for periodontal surgery were excluded from the study

Ages: 19 Years to 52 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2022-03-24 (Actual); Study Completion 2022-03-24 (Actual)

PRIMARY OUTCOMES:
The percentage of Root Coverage (RCP) | Baseline and 6 months
  In this study, the difference between the root surface coverage rate in areas with gingival recession was evaluated by subtracting the 6th month recession depth from the pre-treatment recession depth.
Clinical Attachment Level | baseline and 6th months
  The distance from the mid-buccal point of the teeth to the groove/pocket base based on the cemento-enamel junction was measured in mm with a periodontal probe.
Recession Depth | baseline and 6th month
  The mid-buccal point of the teeth with gingival recession was measured with a periodontal probe, taking the cemento-enamel junction as the basis, until the coronal part of the gingival margin.
Width of Keratinized Tissue | baseline and 6th month
  Clinically, it is determined by subtracting the distance between the free gingival margin and the mucogingival line from the distance to the groove/pocket base.
Transgingival Gingival Thickness | baseline and 6th month
  In this study, gingival thickness was determined by the transgingival probing method.
Gingival İndex | Baseline and 6th month
  Loe ve Silness, 1963 (0-3, skor)
Plaque Index | baseline and 6th month
  Silness ve Löe, 1966
Probing Depth | baseline and 6th month
  Each tooth was measured from the gingival margin to the sulcus base using a periodontal Williams probe, and probing depths were recorded.

SECONDARY OUTCOMES:
Oral Health Impact Profile-14 and Provoked Sensitivity (PS), | baseline and 6th month
  Postoperative morbidity was assessed using quality of life measurements (Oral Health Impact Profile-14, OHIP-14), provoked sensitivity (PS), and the operation durations of the groups. PS was evaluated preoperatively at the recession sites to detect dentin hypersensitivity by applying a 3-second air spray provocation administered by the clinician.

CONTACTS AND LOCATIONS:
Overall Officials: Nazlı Z ALPASLAN, Principal Investigator — Ankara Yildirim Beyazit University, Faculty of Dentistry
Locations (1):
- Van Yuzuncu Yıl University, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bakhishov H, Isler SC, Bozyel B, Yildirim B, Tekindal MA, Ozdemir B. De-epithelialized gingival graft versus subepithelial connective tissue graft in the treatment of multiple adjacent gingival recessions using the tunnel technique: 1-year results of a randomized clinical trial. J Clin Periodontol. 2021 Jul;48(7):970-983. doi: 10.1111/jcpe.13452. Epub 2021 Apr 7. PMID 33751615